CLINICAL TRIAL: NCT00698789
Title: A Double-blind, Placebo Controlled, Randomized Study to Evaluate the Safety and Tolerability of INCB019602 Plus Metformin Compared to Metformin Alone in Type 2 Diabetic Subjects
Brief Title: Evaluate the Safety and Tolerability of INCB019602 When Administered With Metformin in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ended after diabetes development plan review. .
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 19602-201
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A (Experimental): 5 mg of INCB019602 in AM with placebo administration in PM
  Interventions: Drug: INCB019602; Drug: Placebo; Drug: Metformin
- Treatment B (Experimental): 20 mg of INCB019602 in AM with placebo administration in PM
  Interventions: Drug: INCB019602; Drug: Placebo; Drug: Metformin
- Treatment C (Experimental): 5 mg of INCB019602 in PM with placebo administration in AM
  Interventions: Drug: INCB019602; Drug: Placebo; Drug: Metformin
- Treatment D (Experimental): 20 mg of INCB019602 in PM with placebo administration in AM
  Interventions: Drug: INCB019602; Drug: Placebo; Drug: Metformin
- Treatment E (Experimental): 7.5 mg of INCB019602 in PM QoD with placebo administration in AM as well as PM on non active dose days
  Interventions: Drug: INCB019602; Drug: Placebo; Drug: Metformin
- Treatment F (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: INCB019602 — 5 mg of INCB019602 in AM with placebo administration in PM
  Arms: Treatment A
Drug: INCB019602 — 20 mg in AM with placebo administration in PM
  Arms: Treatment B
Drug: INCB019602 — 5 mg in PM with placebo administration in AM
  Arms: Treatment C
Drug: INCB019602 — 20 mg in PM with placebo administration in AM
  Arms: Treatment D
Drug: INCB019602 — 7.5 mg in PM QoD with placebo administration in AM as well as PM on non-active dose days
  Arms: Treatment E
Drug: Placebo — Placebo administration in AM or PM depending on treatment arm dosing regimen.
Drug: Metformin — Stable dose metformin monotherapy

SUMMARY:
Determine the effect of treatment with INCB019602 administered as an add-on to stable dose metformin therapy in type 2 diabetic subjects on safety and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of T2D
* Currently taking metformin monotherapy at a stable dose level
* FPG between 150 and 270 mg/dL

Exclusion Criteria:

* History or clinical manifestations of renal impairment
* Hyperglycemia > 270 mg/dL
* Receiving thiazolidenediones, Exenatide or sulfonylureas within 90 days prior to screening
* Prior use of Acipimox which is known under the name Olbetam within 90 days prior to screening.
* Diagnosed major depression within the last 2 years requiring hospitalization
* History of chronic insulin therapy for glycemic control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by monitoring of AEs, vital signs, ECGs, physical examinations, and clinical laboratory blood and urine parameters. | End of Study

SECONDARY OUTCOMES:
Change from Baseline in fasting plasma glucose and population pharmacokinetics of INCB019602 in type 2 diabetic patients. | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: William V Williams, MD, Study Director — Incyte Corporation
Locations (22):
- United States (22):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Chula Vista, California
  - Los Angeles, California
  - Mission Viejo, California
  - Orange, California
  - Paramount, California
  - San Diego, California
  - Santa Ana, California
  - Tustin, California
  - Colorado Springs, Colorado
  - St. Petersburg, Florida
  - Shawnee Mission, Kansas
  - Shreveport, Louisiana
  - Dearborn, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Elizabeth, New Jersey
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - East Providence, Rhode Island
  - San Antonio, Texas